CLINICAL TRIAL: NCT05864729
Title: Correlation Between Physiological Measures of Ischemia in the Hemodynamics Laboratory and Systemic Microcirculatory Parameters in Patients With Intermediate Lesions of the Main Coronary Arteries
Brief Title: The Association Between Systemic Microvascular Endothelial Function and Coronary Physiology Indexes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Principal Investigator, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAE: 28368620.7.0000.5272
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Myocardial Ischemia
Keywords: endothelial function; coronary flow reserve; laser speckle
MeSH Terms: conditions — Myocardial Ischemia | interventions — Coronary Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary angiography with physiological lesion assessment by fractional flow reserve (FFR) and contrast fractional flow reserve (cFFR). — Hemodynamic invasive study employing FFR (after intracoronary adenosine administration) and cFFR (after intracoronary lopamidol contrast media administration) measurements of hyperemic intravascular pressure.
  Other Names: Evaluation of systemic skin microvascular endothelial function

SUMMARY:
The present study evaluates skin microvascular reactivity and coronary physiology in the same coronary artery disease (CAD) patients.

This study is expected to find associations between systemic microvascular reactivity, measured non-invasively at the skin surface, and coronary reserve evaluated by the invasive angiographic method.

DETAILED DESCRIPTION:
Introduction: Microvascular reactivity (MR) evaluated in the skin has been proposed as representative of systemic endothelial function, including coronary circulation. There is a lack of studies investigating the association between skin MR and invasive evaluation of coronary reserve. Objective: To evaluate skin MR and coronary physiology in the same coronary artery disease (CAD) patients. Methods: Transversal study, recruiting adult patients with indication for elective coronary angiographic study for the evaluation of CAD by an independent medical team. The evaluation of microvascular cutaneous blood flow of the forearm will use laser speckle contrast imaging (LSCI) coupled with acetylcholine iontophoresis. Coronary physiology will be evaluated in the same patients and in the same day with coronary angiography with lesion assessment by fractional flow reserve (FFR, after intracoronary adenosine administration) and contrast fractional flow reserve (cFFR, after intracoronary contrast media administration), with measurements of hyperemic intravascular pressures. FFR and cFFR will be performed in vessels with intermediate lesions, as evaluated in quantitative angiography. Expected results: This study is expected to find associations between systemic MR, measured non-invasively at the skin surface, and coronary reserve evaluated by the invasive angiographic method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermediate obstructive coronary artery disease (40-80% lumen obstruction of epicardial vessels or 30-60% obstruction of left main coronary artery).

Exclusion Criteria:

* ST elevation myocardial infarction in the first 72 hours of evolution.
* Allergy to contrast media or adenosine
* Asthma or chronic obstructive pulmonary artery disease diagnosis
* Ongoing acute coronary syndrome
* Systolic blood pressure under 90mmHg
* Baseline arrhythmias or advanced atrioventricular blockade
* Advanced arterial calcification
* Renal failure (defined as serum creatinine above 1.5mg/dl)
* Saphenous graft or mammary artery graft anastomosis stenosis
* Severe left ventricular systolic dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment by fractional flow reserve (FFR) and contrast fractional flow reserve (cFFR). | day 1 visit to the hemodynamic laboratory
  Physiological coronary artery obstruction assessment through FFR and cFFR. For FFR and cFFR measurement, a 0.014FR guidewire will be advanced distal to the lesion, with baseline and hyperemic (after adenosine or contrast administration) vascular pressure measurements, with two-minute interval between each measurement.

SECONDARY OUTCOMES:
Systemic microvascular reactivity | day 1 visit to the hemodynamic laboratory
  Laser-based method for evaluating non-invasive, operator-independent systemic microvascular function that detects microvascular flow in the skin for the evaluation of systemic vascular endothelial function.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No